CLINICAL TRIAL: NCT03607760
Title: Extracorporeal Membrane Oxygenation (ECMO) and Neonatal Outcomes:a Retrospective Multicenters Study
Brief Title: Extracorporeal Membrane Oxygenation (ECMO)
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Bayi Children's Hospital Affiliated to PLA Army General Hospital, China (Other); Children's Hospital of Chongqing Medical University (Other); Hunan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Beijing 302 Hospital (Other); Navy General Hospital, Beijing (Other); Zhengzhou Children's Hospital, China (Other); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: ECMO
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2018-11

CONDITIONS: Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO: severe respiratory failure with ECMO
  Interventions: Device: ECMO
- conventional mechanical ventilation: severe respiratory failure with conventional mechanical ventilation
  Interventions: Device: conventional mechanical ventilation

INTERVENTIONS:
Device: ECMO — the patients with severe respiratory failure were supported by ECMO
  Groups: ECMO
Device: conventional mechanical ventilation — the patients with severe respiratory failure were supported by conventional mechanical ventilation
  Groups: conventional mechanical ventilation

SUMMARY:
Since the 1970s, extracorporeal membrane oxygenation (ECMO) support has been used to support gas exchange for children with severe acute respiratory failure who fail mechanical ventilation. ECMO is more expensive than each of these other procedures.But its action is unclear

DETAILED DESCRIPTION:
Since 1974, eight randomized controlled trials have been reported in ECMO for respiratory failure, and none have included non-neonatal pediatric patients. Cochrane systematic reviews of this evidence concluded that ECMO for neonatal respiratory failure had a survival advantage, but there was insufficient evidence to demonstrate a survival advantage for ECMO used to support respiratory failure in adults. Moreover, these trials were performed prior to 2009, and since then advances in ECMO technology have enhanced the delivery of ECMO support, and new research has changed conventional management of severe acute respiratory distress syndrome (ARDS)

ELIGIBILITY:
Inclusion Criteria:

1. ECMO group:

1. Oxygenation Index > 40 for >4 hours
2. Failure to wean from 100% oxygen despite prolonged (> 48h) maximal medical therapy or persistent episodes of decompensation
3. Severe hypoxic respiratory failure with acute decompensation (PaO2 <40) unresponsive to intervention
4. Severe pulmonary hypertension with evidence of right ventricular dysfunction and/or left ventricular dysfunction. The pulmonary artery pressure > 60mmHg evaluated by the Echo, arterial duct keeps open and the blood flow was either by-level shunt or completely shunt from right side to left side.

2. Non-ECMO group:

1. Oxygenation Index > 16 and reach the Montreux definition of severe respiratory distress syndrome
2. Vasoactive-inotropic score (VIS) ≥ 40 [VIS=dopamine dose (μg/kg/min)×1 + dobutamine dose (μg/kg/min)×1 + milrinone dose (μg/kg/min)×10 + amrinone dose (μg/kg/min)×10 + epinephrine dose (μg/kg/min)×100 + isoprenaline dose (μg/kg/min)×100]

Exclusion Criteria:

1. Gestational age < 36 weeks, birth weight < 2 kg, day post-birth > 28 days.
2. lethal chromosomal disorder (includes trisomy 13, 18 but not 21) or any other lethal anomaly
3. irreversible brain damage
4. uncontrolled bleeding
5. Grade III or greater intraventricular hemorrhage
6. ventilator days ≥ 15 days.

Ages: 1 Hour to 1 Month | Sex: All
Age Groups: Child
Study Population: All the patients will be eligible only when they reach the cutting line in the following:
  Gestational age > 36 weeks, birth weight > 2 kg, day post-birth < 28 days.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | 36 weeks' gestational age or before discharge from hospital
  the patients died
28 days' mortality | 28 days
  the patients died

SECONDARY OUTCOMES:
Neonatal necrotizing enterocolitis | 36 weeks' gestational age or before discharge from hospital
  Neonatal necrotizing enterocolitis was diagnosed after extubation
Intraventricular hemorrhage | 36 weeks' gestational age or before discharge from hospital
  Intraventricular hemorrhage was diagnosed after extubation
bronchopulmonary dysplasia | 36 weeks' gestational age or before discharge from hospital
  bronchopulmonary dysplasia was diagnosed after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China